CLINICAL TRIAL: NCT04515121
Title: Effects of High-definition Transcranial Electrical Stimulation on the Lower Extremity in Patients With Stroke
Brief Title: High-definition Transcranial Electrical Stimulation for Lower Limb Stroke Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Principal Investigator, Lai chien hung, Professor, Taipei Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N202004091
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Stroke
Keywords: Stroke, Transcranial electrical stimulation, Lower-limb rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HD-tCES & lower limb rehabilitation (Experimental): The experiment group will receive HD-tCES combined with lower limb rehabilitation of affected side.
  Interventions: Device: HD-tCES; Other: Lower limb rehabilitation
- Sham HD-tCES & lower limb rehabilitation (Sham Comparator): The sham control group will receive sham HD-tCES combined with lower limb rehabilitation of affected side.
  Interventions: Device: Sham HD-tCES; Other: Lower limb rehabilitation

INTERVENTIONS:
Device: HD-tCES — The high definition transcranial electrical stimulation was applied using a 1*4 ring electrode configuration. The anodal electrode was placed on the ipsilesional C1/C2, and the remaining 4 cathodal electrodes were placed in a radius of approximately 7.5 cm from anode (Cz, F3, T7, and P3 on the left hemisphere or Cz, F4, T8, and P4 on the right hemisphere). HD-tCES will be applied for 20 minutes at an intensity of 1.0 mA direct current stimulation and a specific-added waveform each time, 3 times a week, lasting for 4 weeks.
  Arms: HD-tCES & lower limb rehabilitation
Device: Sham HD-tCES — The high definition transcranial electrical stimulation was applied using a 1*4 ring electrode configuration. The anodal electrode was placed on the ipsilesional C1/C2, and the remaining 4 cathodal electrodes were placed in a radius of approximately 7.5 cm from anode (Cz, F3, T7, and P3 on the left hemisphere or Cz, F4, T8, and P4 on the right hemisphere). Sham HD-tCES will consist of a 5-second ramp up to 1.0 mA direct current stimulation and a specific-added waveform followed immediately by a 5-second ramp down, no current in the middle 19 minutes 40 seconds, and a ramp-up and ramp-down period during the last 10 seconds.
  Arms: Sham HD-tCES & lower limb rehabilitation
Other: Lower limb rehabilitation — Lower limb rehabilitation programs will be selected and graded in accordance with each patient's lower limb function and specific aims of activities of daily living. Lower limb rehabilitation will be provided for 30 minutes each time, 3 times a week, lasting for 4 weeks.

SUMMARY:
Transcranial electrical stimulation (tCES) is a non-invasive and safe treatment, which uses a low direct current or alternating current to change the excitability of the cerebral cortex. The tCES has been applied in clinical trials related to rehabilitation research in recent years, and the safety and effectiveness have also been established. However, the existing tCES products effect on the whole brain networks and lack special waveforms. We developed a wearable high-definition tCES (HD-tCES) with special waveforms. This novel stimulation system will result in more precise and focal stimulation of selected brain regions with special waveforms to display better neuromodulation performance. In this study, we will preliminarily examine the effects and safety of the HD-tCES on lower extremity in patients with stroke. We expect that the HD-tCES combined with the lower extremity rehabilitation can shorten the duration of rehabilitative periods, improve stroke patients' activity of daily living, reduce the care burden of patients' family, and subsequently decrease the cost of health care insurance.

ELIGIBILITY:
Inclusion Criteria:

1. With a diagnosis of stroke.
2. Age ≥ 20 years.
3. Hemiplegia, Brunnstrom stage III-V.
4. 6 months to 5 years after stroke.
5. Muscular inelasticity (spasticity) 1-3 on the affected lower limb, evaluated by the Modified Ashworth Scale.
6. Ability to walk for 10 min non-stop with no gait aids or ability to walk 20 m with supervision or slight assistance.

Exclusion Criteria:

1. Intolerance to electrical stimulation.
2. Contracture on lower extremities, and limitation in joint range of motion.
3. Severe spasticity.
4. Ossification or inflammation in muscle tissue.
5. A history of arrhythmia.
6. Implantable medical electronic devices (e.g., like pacemaker).
7. Metal implants in the head or neck.
8. Wounds on the skin of head.
9. A history of brain surgery or severe brain trauma.
10. Severe cognitive or psychiatric disorders (e.g., schizophrenia, depression or bipolar disorder).
11. A history of seizure or other brain pathology.
12. Drug or alcohol abuse.
13. Malignant neoplasm or rheumatism disorder (e.g., SLE, RA, AS, IBD)
14. Undergoing other non-invasive brain stimulation.
15. Intra-cerebral lesions (such as brain tumors, arteriovenous tumors).
16. History of encephalitis or meningitis.
17. Stroke lesion in cerebellum or brainstem.
18. Leg amputation.
19. Sleep deprivation.
20. Severe or recent heart disease.
21. Subjects who use drugs that may lower the seizure threshold.
22. Pregnant or breastfeeding women.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-08-20 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Fugl-Meyer Assessment lower extremity scale (FMA-LE) after intervention | Baseline (within 7 days ahead to the 1st intervention session) and after 4-week intervention (within 7 days after the last intervention session)
  The FMA-LE assesses motor functioning of lower extremity. Each movement is estimated by a 3-point scale (0-1-2). The total score of the FMA-LE is 34, and a higher score indicates that the patient has better movement ability.

SECONDARY OUTCOMES:
Change from baseline in the Berg Balance Scale (BBS) after intervention | Baseline (within 7 days ahead to the 1st intervention session) and after 4-week intervention (within 7 days after the last intervention session)
  The BBS is used to objectively determine a patient's ability to safely balance during a series of predetermined tasks. It contains 14 items with each item consisting of a five-point ordinal scale ranging from 0 to 4. A higher score indicates that the patient has better balance.
Change from baseline in the Timed Up and Go Test (TUG) after intervention | Baseline (within 7 days ahead to the 1st intervention session) and after 4-week intervention (within 7 days after the last intervention session)
  The TUG assesses a patient's mobility and requires both static and dynamic balance. It measures the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.
Change from baseline in the Gait Evaluation after intervention | Baseline (within 7 days ahead to the 1st intervention session) and after 4-week intervention (within 7 days after the last intervention session)
  The Gait Evaluation includes cadence, stride duration, stride length, and velocity.
Change from baseline in the Modified Ashworth Scale (MAS) after intervention | Baseline (within 7 days ahead to the 1st intervention session) and after 4-week intervention (within 7 days after the last intervention session)
  The MAS is commonly used in clinical practice for grading spasticity. The MAS is rated on a 6-point scale (0, 1, 1+, 2, 3, 4), and a higher score indicates that the patient has higher muscle tension. The muscles being assessed include hip flexor, hip extensor, knee flexor, knee extensor, ankle dorsiflexor, and ankle plantarflexor.
Change from baseline motor evoked potential (MEP) after intervention | Baseline (within 7 days ahead to the 1st intervention session) and after 4-week intervention (within 7 days after the last intervention session)
  The MEP elicited in peripheral muscles by transcranial magnetic stimulation over motor cortex is one of the hallmark measures for non-invasive quantification of cortical excitability.
Incidence of treatment-emergent adverse events | Within 10 minutes after each intervention session (a total of 12 sessions, 3 sessions/week, lasting 4 weeks)
  Immediately after each HD-tCES stimulation, the patient will be questioned about eventual side effect.

CONTACTS AND LOCATIONS:
Locations (3):
- Taiwan (3):
  - Taipei Medical University-Shuang Ho Hospital,Ministry of Health and Welfare, New Taipei City
  - Taipei Medical University Hospital, Taipei
  - Taipei Municipal Wanfang Hospital - Taipei Medical University, Taipei

IPD SHARING:
Plan to Share IPD: No